CLINICAL TRIAL: NCT00226421
Title: An Open-Label Titration Followed by a Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Tolerability, and Safety of Oxymorphone Extended Release Tablets in Opioid-Experienced Patients With Chronic Low Back Pain
Brief Title: Efficacy and Safety of Oxymorphone Extended Release in Opioid-Experienced Patients With Chronic Non-Malignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director Clinical R&D
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3202-032
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pain
Keywords: opioid; oxymorphone; chronic pain; randomized, double-blind trial; low back pain
MeSH Terms: conditions — Chronic Pain; Low Back Pain

INTERVENTIONS:
Drug: Oxymorphone Extended Release

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy and safety of oxymorphone extended release in opioid-experienced patients with chronic low back pain.

DETAILED DESCRIPTION:
Patients with chronic low back pain on stable opioid treatment will be converted to oxymorphone extended release (ER)and enter an open-label treatment phase.During the Open-Label Titration Period (up to 28 days), patients will receive daily oxymorphone ER PO q12h. Patients stabilized on a dose that provides adequate pain relief will be randomized to either continue on the stabilized dose of oxymorphone ER or receive placebo in a double-blind fashion for a total duration of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older
* In good health as determined by the Investigator on the basis of medical history and physical examination.
* Moderate to severe chronic non-neuropathic low back pain that has been present daily for at least several hours per day for a minimum of three months prior to the screening.
* On a stable around-the-clock opioid pain medication for the management of moderate to severe chronic lower back pain.
* Expected to require a total daily oxymorphone ER dose that is a minimum of 20 mg per day (oral morphine equivalent: approximately 60 mg) and will not exceed 220 mg oxymorphone ER (oral morphine requirement: approximately 660 mg).
* Any adjunct therapy for back pain such as physical therapy, biofeedback therapy, acupuncture therapy or herbal remedies, based on the patient's current status should remain unchanged during the period of participation of the patient.
* Written informed consent

Exclusion Criteria:

* Pregnant and/or lactating
* Subjects with radiculopathy, fibromyalgia, reflex sympathetic dystrophy or causalgia (complex regional pain syndrome), acute spinal cord compression, cauda equina compression, acute nerve root compression, severe lower extremity weakness or numbness, bowel or bladder dysfunction secondary to cauda equina compression, diabetic amyotrophy, meningitis, discitis, or back pain due to secondary infection or tumor.
* Cannot or will not agree to stop local regional pain treatments during the study (nerve/plexus blocks or ablation, neurosurgical procedures for pain control, Botulinum toxin injections, or inhalation analgesia). The patient must not have a nerve/plexus block within 4 weeks of screening (Visit 1). The patient must not have a Botulinum toxin injection in the lower back region within 3 months of screening.
* Intend to alter their physical therapy regimen during the study.
* Surgical procedures directed towards the source of back pain within 6 months of screening.
* Pain which is secondary to confirmed or suspected neoplasm.
* Dysphagia or difficulty swallowing tablets or capsules.
* Significant prior history of substance abuse or alcohol abuse.
* Use of any investigational medication within 30 days prior to the first dose of study medication.
* Previous exposure to oxymorphone.
* History of clinically significant intolerance to oxymorphone or a known hypersensitivity to opioid analgesics.
* History of seizure.
* use of MAO inhibitor within 14 days prior to the start of study medication.
* Other clinically significant conditions as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-10; Study Completion 2005-08

PRIMARY OUTCOMES:
Change in pain intensity from baseline (pre-randomization) to last assessment.

SECONDARY OUTCOMES:
- Time to early discontinuation due to lack of efficacy
- Patient's Global Assessment of Pain Medication
- Physician's Global Assessment of Pain Medication
- Pain Quality Assessment Scale
- Safety as measured by AEs

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Southern Drug Research, Hueytown, Alabama
  - Phoenix Center for Clinical Research, Phoenix, Arizona
  - Arizona Research, Phoenix, Arizona
  - Express Care Clinical Research, Colorado Springs, Colorado
  - Glasgow Family Practice, Newark, Delaware
  - Radiant Research, Daytona Beach, Florida
  - University Clinical Research, DeLand, Florida
  - LCFP Inc., Fort Myers, Florida
  - Century Clinical Research, Holly Hill, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Radiant Research, Pinellas Park, Florida
  - Park Place Therapeutic Center, Plantation, Florida
  - Comprehensive Neurology Specialists, Atlanta, Georgia
  - Comprehensive Neuroscience, Atlanta, Georgia
  - Pain Specialists of Greater Chicago, Burr Ridge, Illinois
  - Mid-America Physiatrists, Overland Park, Kansas
  - Research Medical Center, Kansas City, Missouri
  - Radiant Research, St Louis, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Piedmont Anesthesia, Winston-Salem, North Carolina
  - Health Research Institute, Oklahoma City, Oklahoma
  - Pain Consultants of Oregon, Eugene, Oregon
  - Keystone Medical Research, Altoona, Pennsylvania
  - Perkiomen Valley Family Practice, Collegeville, Pennsylvania
  - Feasterville Family Health Center, Feasterville, Pennsylvania
  - Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Paragon Clinical Research, Cranston, Rhode Island
  - Waccamaw Pain Management, Murrells Inlet, South Carolina
  - KRK Medical Research, Richardson, Texas
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Peniston JH, Hu X, Potts SL, Wieman MS, Turk DC. Tolerability of concomitant use of selective serotonin reuptake inhibitors or serotonin-norepinephrine reuptake inhibitors and oxymorphone extended release. Postgrad Med. 2012 Mar;124(2):114-22. doi: 10.3810/pgm.2012.03.2542. PMID 22437221
- [Derived] Peniston JH, Xiang Q, Gould EM. Factors affecting acceptability of titrated oxymorphone extended release in chronic low back pain - an individual patient analysis. Curr Med Res Opin. 2010 Aug;26(8):1861-71. doi: 10.1185/03007995.2010.490457. PMID 20521870